CLINICAL TRIAL: NCT05655325
Title: Accelerated Age-related Cognitive Decline: Impact of Exercise on Executive Function and Neuroplasticity
Acronym: EXEC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Ulf Bronas, Professor of Biobehavioral Science (in Nursing), Columbia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AAAU9751; 2022-0311 (Other: UIC); R01AG076456 (NIH)
Record Dates: First submitted 2022-12-01; First posted 2022-12-19 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Mild Cognitive Impairment; Chronic Kidney Diseases
Keywords: mild cognitive impairment; chronic kidney disease; exercise; Lifestyle behavior; home-based exercise
MeSH Terms: conditions — Cognitive Dysfunction; Renal Insufficiency, Chronic; Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial. Participants are randomized following baseline testing using block randomization of 2 and 4 to either an exercise intervention group or a health education group
Who Masked: Investigator, Outcomes Assessor
Masking Description: The PI and the outcome assessors are blinded to group assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Home-based walking exercise (Experimental): A 6-month partially supervised walking exercise training using a tapered approach. Participants begin with exercising (walking) in person, on-site one time per week and 3 times per week at home for a minimum exercise dosage of 30 minutes of accumulated exercise per session during month 1. During month 2, participants will exercise on-site once every other week and 3-4 times per week at home a minimum exercise dosage of 30 minutes of accumulated exercise per session. During months 2-6, participants will exercise at home 4 times per week for a minimum exercise dosage of 30 minutes of accumulated exercise per session and they will receive a phone call every two weeks to help coach and address any problems. Participants will receive a Fitbit fitness tracker that will be used to deliver their personalized exercise program, exercise monitoring, feedback, and motivational messages.
  Interventions: Behavioral: Home-based walking exercise
- Health education (Placebo Comparator): The health education group will receive the same amount of contact hours as the intervention group. The attention control group will receive health education and stretching exercises. Participants will be in person, on-site one time per week during month 1 for about 30 minutes. During month 2, participants will attend the health education on-site once every other week for about 30 minutes. During months 2-6 participants will receive a phone call every two weeks to help remind about the health education. Participants will receive a Fitbit fitness tracker that will be used for exercise monitoring.
  Interventions: Other: Attention control

INTERVENTIONS:
Behavioral: Home-based walking exercise — A 6-month partially supervised walking exercise program using a tapered approach.Participants will begin exercise (walking) at a relatively low intensity and progress to moderate intensity. Intensity will start at 40% and progress as tolerated up to 60-70%. Rating of perceived exertion of 12-14 (fairly light to moderate) will be used to aid intensity (Rating of perceived exertion 6-20 scale). This is an accepted method for achieving desired exercise intensity. Participants will progress over time to exercise 3-4/week for 30-45 minutes. The exercise program may need to be adjusted for (e.g. 10 minutes of exercise 3 times), to achieve the minimum exercise dose of 30 minutes. This will be determined for each individual participants as needed.
  Arms: Home-based walking exercise
Other: Attention control — Health education and stretching
  Arms: Health education

SUMMARY:
The purpose of this study is to see if 6 months of home-based walking will improve memory, and brain structure and function, compared to health education in older adults that have chronic kidney disease and mild cognitive impairment.

DETAILED DESCRIPTION:
Following informed consent, participants will undergo tests for heart health, physical function, memory testing, and brain structure and function using imaging (taking pictures of the brain with an MRI). Following these tests participants are randomized to a home-based walking program or health education for 6 months. Participants are given a fitness tracker and gets ongoing telephone coaching during the 6 months. After 6 months the tests are repeated.

ELIGIBILITY:
Inclusion Criteria:

* • Diagnosed stage 3-4 chronic kidney disease (CKD, estimated glomerular filtration rate (eGFR) <60 to 20 ml/min);

  * >55 yrs of age
  * Mild cognitive impairment (18-26 on the MOCA)
  * ability to undergo an MR
  * no history of major head trauma (No head trauma/concussion with loss of consciousness)
  * Speaks, reads, writes English

Exclusion Criteria:

* • Diagnosed Dementia or a Clinical Dementia Rating Scale score of <2, or a MOCA of <18

  * Participating in a supervised exercise program with intent to increase fitness levels 3 days/week,
  * Requires assistive ambulation
  * Limited exercise capacity due to claudication; unstable angina, severe arthritis, extreme dyspnea on exertion, unstable coronary artery disease
  * Class III-IV heart failure
  * History of uncontrolled sustained arrhythmias, severe/symptomatic aortic or mitral stenosis, hypertrophic obstructive cardiomyopathy, severe pulmonary hypertension, active myocarditis/pericarditis, thrombophlebitis, and recent systemic/pulmonary embolus
  * Resting systolic BP >200 mmHg or resting diastolic BP >110 mmHg
  * Any unforeseen illness or disability that would preclude cognitive testing or exercise training
  * One or more contraindication for MRI; cardiac pacemaker, aneurysm clip, cochlear implants, shrapnel, history of metal fragments in eyes, neurostimulators, diagnosed claustrophobia (MRI only)
  * Any self-reported major psychiatric disorders requiring medical therapy (e.g. schizophrenia, bipolar disorder).
  * Self-reported new diagnosis of clinical depression within 3 months of enrollment or unstable clinical depression requiring medication adjustment within 3 months of enrollment

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2024-06-18 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in Executive Function from baseline | Change from baseline at 6 months
  Composite score from Phonemic and Semantic Fluency total correct words; Trail Making Test Part B (TMT-B) time to completion; Digit Span subtest backwards total score. The composite executive functioning score will be created by converting these four individual executive cognitive scores (phonemic and Semantic fluency score), digit span backward subtest, and trail making test part B (following directionality conversion)) to standardized z scores and then averaging the standardized z scores. Z-score range from -3 to +3. Higher score is better.
Change in processing speed from baseline | Change from baseline at 6 months
  Trail making test part A (TMT-A) time to completion in seconds. Faster completion is better.
Change in attention/information processing from baseline | Change from baseline at 6 months
  Digit symbol substitution test total number correct. Higher number is better.
Change in Learning and Memory short recall | Change from baseline at 6 months
  California verbal learning test-II, short recall total number of words correct. Higher number is better.
Change in Learning and Memory long recall | Change from baseline at 6 months
  California verbal learning test-II long recall total number of words correct. Higher number is better.
Change in Learning and Memory learning slope | Change from baseline at 6 months
  California verbal learning test-II leaning slope (average number of new words recalled during five consecutive learning trials). Higher number is better.
Change in Learning and Memory recognition memory discrimination | Change from baseline at 6 months
  California verbal learning test-II recognition memory discrimination total number of words correct. Higher number is better.
Change in global cognitive function | Change from Baseline to 6 months
  Composite score from Phonemic and Semantic Fluency total correct words; Trail Making Test Part B time to completion; Digit Span subtest backwards total score; Digit symbol substitution test total correct and trail making test part A time to completion; California verbal learning test-II, short and long recall, leaning slope, recognition memory discrimination total correct. The composite global cognitive score will be created by converting these 10 individual cognitive scores (following directionality change of TMT-A and TMT-B) to standardized z scores and then averaging the standardized z scores. Z score range from -3 to +3. Higher score is better.

SECONDARY OUTCOMES:
Change from baseline to 6-months in white matter fractional anisotropy. | Change from baseline to 6 months
  Quantify change from baseline to 6-months in white matter integrity fractional anisotropy using diffusion tensor MRI imaging. Range 0-1. Higher number is better.
Change from baseline to 6-months in white matter mean diffusivity. | Change from baseline to 6 months
  Quantify change from baseline to 6-months in white matter integrity mean diffusivity using diffusion tensor MRI imaging. Range 0-1. Lower number is better.
Changes from baseline to 6-months in functional connectivity | Change from Baseline to 6 months
  Quantify change from baseline to 6-months in functional connectivity using functional MRI (fMRI). Range 0-1. Higher score is better.
Change from baseline to 6-months in cerebral blood flow. | Change from baseline to 6 months
  Quantify changes from baseline to 6-months in cerebral blood flow using perfusion MRI arterial spin labeling in mL/100g/min. Higher is better.
Change from baseline to 6-months in hippocampal volume | Change from baseline to 6 months
  Quantify change from baseline to 6-months in hippocampal volume using morphometry using 3D T1-weighted MRI in milliliters cubed. Higher number is better.

CONTACTS AND LOCATIONS:
Overall Officials: Ulf G Bronas, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be made available based on each publication. The PI will share data through sharing requests. All data will be properly de-identified before sharing. Data sharing requests may be granted to those that 1) have a detailed research plan for the requested data, 2) have human subjects training, and 3) have institutional review board (IRB) approval from their home institution. Data sharing requests will be furnished with a data-sharing agreement approved by the University of Illinois Chicago IRB that contains commitments to: 1) Using the data for research purposes only (no commercial use of the data), 2) not attempting to re-identify any participant, 3) securing the data using appropriate technology, and 4) destroying or returning the data after analyses. Other stipulations may be added to the data-sharing agreement if deemed necessary. Data may be shared as a complete or partial dataset depending on the request.
Supporting Information: Study Protocol, SAP
Time Frame: IPD will be made available by the time of online publication based on each manuscript. Data will be available for 10 years.
Access Criteria: PI will share data through sharing requests and also work with the Program Officer to identify relevant NIH-approved and University of Illinois Chicago data repositories for the data.Data sharing requests may be granted to those that 1) have a detailed research plan for the requested data, 2) have human subjects training, and 3) have IRB approval from their home institution. Data sharing requests will be furnished with a data-sharing agreement approved by the University of Illinois Chicago IRB that contains commitments to: 1) Using the data for research purposes only (no commercial use of the data), 2) not attempting to re-identify any participant, 3) securing the data using appropriate technology, and 4) destroying or returning the data after analyses. Other stipulations may be added to the data-sharing agreement if deemed necessary. Data may be shared as a complete or partial dataset depending on the request.